CLINICAL TRIAL: NCT00997399
Title: A Phase I, Open-label, Multi-center Study to Evaluate the Pharmacokinetics and Safety of Oral Panobinostat in Patients With Advanced Solid Tumors and Varying Degrees of Renal Function
Brief Title: Study to Evaluate Panobinostat (DACi) Pharmacokinetics and Safety in Solid Tumors and Varying Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLBH589X2105; 2009-012263-34 (EudraCT Number)
Record Dates: First submitted 2009-10-15; First posted 2009-10-19 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2019-07

CONDITIONS: Advanced Solid Tumors
Keywords: Ph I; panobinostat (DACi); PK & safety; solid tumors; varying renal function; advanced
MeSH Terms: interventions — Panobinostat

ARMS (1):
- LBH589 (Experimental)
  Interventions: Drug: panobinostat (LBH589)

INTERVENTIONS:
Drug: panobinostat (LBH589)

SUMMARY:
Panobinostat (LBH589) is a deacetylase inhibitor (DACi) which belongs to a structurally novel cinnamic hydroxamic acid class of compounds. It is one of the most potent class I/II pan-DAC inhibitor (pan-DACi) that has shown anti-tumor activity in pre-clinical models and patients with solid tumors and hematological malignancies.

To date, the pharmacokinetics (PK) of panobinostat has been characterized in patients with solid tumors and hematological malignancies participating in several phase I/II clinical studies. Panobinostat PK does not appear to be different in patients with solid tumors and hematological malignancies. However, the effect of organ dysfunction on PK of panobinostat is yet to be elucidated.

Kidney and liver are involved in the elimination and metabolism of panobinostat. The current study is designed to evaluate the impact of renal function status on panobinostat PK.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has documented diagnosis of advanced solid tumor for which no standard systemic therapy exists
2. Patient has normal or abnormal renal organ function
3. Patient has provided written informed consent prior to any screening procedures

Exclusion Criteria:

1. Patient needing valproic acid for any medical condition during the study or within 5 days prior to the first panobinostat dose
2. Patient received prior treatment with DAC inhibitors including panobinostat
3. Patient requiring dialysis
4. Patient requiring diuretics unless patient is taking potassium sparring diuretics
5. Patient has acute renal failure, history of transplant, ESRD (however acceptable severe renal impaired group)
6. Female patient who is pregnant or breast feeding or with childbearing potential and not willing to use a double method of contraception up to 3 months after the end of study treatment. Male patient who is not willing to use a barrier method of contraception up to 3 months after the end of study treatment.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To assess the effect of varying degrees of renal function as defined by creatinine clearance), on the pharmacokinetics of panobinostat. | First 7 days

SECONDARY OUTCOMES:
To assess the effect of varying degrees of renal function on the safety of panobinostat | Entire duration of study
To evaluate whether there is a relationship between PK and safety parameters in patients with varying degrees of renal function. | 7 days
To explore anti-tumor activity associated with panobinostat. | 6 months (6 cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- University of Utah / Huntsman Cancer Institute, Salt Lake City, Utah, United States
- Netherlands (2):
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, Utrecht
- Novartis Investigative Site, Sankt Gallen, Switzerland
- Novartis Investigative Site, Merseyside, United Kingdom

REFERENCES:
- [Derived] Sharma S, Witteveen PO, Lolkema MP, Hess D, Gelderblom H, Hussain SA, Porro MG, Waldron E, Valera SZ, Mu S. A phase I, open-label, multicenter study to evaluate the pharmacokinetics and safety of oral panobinostat in patients with advanced solid tumors and varying degrees of renal function. Cancer Chemother Pharmacol. 2015 Jan;75(1):87-95. doi: 10.1007/s00280-014-2612-8. Epub 2014 Nov 7. PMID 25377157
- See also: Results for CLBH589X2105 on the Novartis Clinical Trial Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13704